CLINICAL TRIAL: NCT04490941
Title: The Effectiveness of Ophthalmologist-delivered Health Education on Top of Routine Community Care in Type 2 Diabetic Patients at Risk for Diabetic Retinopathy: A Parallel-group, Randomised Trial
Brief Title: A Trial on Ophthalmologist-delivered Health Education on Top of Routine Community Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SYSU-OPH-007
Record Dates: First submitted 2020-07-22; First posted 2020-07-29 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Ophthalmologist-delivered health education
- Control group (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Ophthalmologist-delivered health education — The educational intervention will be conducted on-site by a qualified, experienced ophthalmologist at an ophthalmic center with goals of building awareness on diabetes symptoms, particularly on diabetic retinopathy, and its risk factors with appropriate management.
  Arms: Intervention group
Other: Usual care — Usual care follows standard procedure on diabetes management similar to the routine service provision.
  Arms: Control group

SUMMARY:
Diabetic retinopathy affects over one third of all people with diabetes and is one of the leading causes of vision loss. The management of diabetes and its complications should include screening for diabetic retinopathy. A randomised trial is therefore needed of the use of a simple and widely practicable approach to explore the integration of eye care in managing diabetes. The trial is designed as a randomised, controlled, superiority trial. The aim is to explore the effectiveness of ophthalmologist-delivered health education on top of routine community care on blood glucose and eye-related clinical outcomes in type 2 diabetic patients at risk for diabetic retinopathy.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is a highly specific vascular complication of diabetes mellitus, with prevalence strongly related to a number of risk factors including the duration of diabetes, the level of glycaemic control, etc. Diabetic retinopathy affects over one third of all people with diabetes and is one of the leading causes of vision loss. It is recommended that optimising glycaemic control could reduce the risk or slow the progression of diabetic retinopathy, and that the management of diabetes and its complications should include screening for diabetic retinopathy. A randomised trial is therefore needed of the use of a simple and widely practicable approach to explore the integration of eye care in managing diabetes. The trial is designed as a randomised, controlled, superiority trial. The aim is to explore the effectiveness of ophthalmologist-delivered health education on top of routine community care on blood glucose and eye-related clinical outcomes in type 2 diabetic patients at risk for diabetic retinopathy. Participants will be randomly assigned to either control or intervention group with a 1:1 allocation as per computer-generated random numbers. A senior onsite manager will monitor participant enrolment over the course of the study. An ophthalmologist-delivered health education will be offered as the intervention in an individualised, face-to-face counselling session to build awareness on diabetes symptoms, particularly on diabetic retinopathy, and its risk factors with appropriate management. All subjects, regardless of the group allocation, will be followed up for 12 months. Baseline and follow-up profiles will be assessed and collected by clinical personnel blind to group allocation. The intervention arm will be compared against the control for all primary analysis. The study was partly supported by the Open Research Funds of the State Key Laboratory of Ophthalmology. Trial results will be disseminated to key stakeholders and the general medical community.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-80 years
* Clinically diagnosed with type 2 diabetes
* At risk of diabetic retinopathy (DR),e.g. no apparent DR or mild non-proliferative DR
* On regular community care by 'family doctor team' in the context of the National basic public health service delivery

Exclusion Criteria:

* With symptoms of cognitive dysfunction, dementia, severe mental disorders, or other conditions with inability to appropriately convey personal thoughts
* Type 1 diabetes or gestational diabetes
* Developed with eye conditions requiring timely treatment, e.g., diabetic macular edema, severe non-proliferative diabetic retinopathy, or proliferative DR
* Have a family member (including relatives) who participated in the trial with a different group assignment
* Currently enrol in other ongoing interventions that may exert additional effects on blood glucose control

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | 12-months follow-up
  Proportion of participants who had optimal control of HbA1c level at 12 months

SECONDARY OUTCOMES:
Treatment burden | 12-months follow-up
  Use of treatment burden questionnaire to quantify item scores for each domain, in detail and together, on treatment burden of patients
Patients' adherence | 12-months follow-up
  Use of adherence questionnaire to examine the extent to which physician advice, in detail and together, are adhered to by patients
Body mass index | 12-months follow-up
  Use of weight and height to report body mass index in kg/m^2
Blood pressure | 12-months follow-up
  Use of systolic and diastolic blood pressure to report blood pressure profile in mmHg
cholesterol concentration | 12-months follow-up
  Use of cholesterol concentration to report lipid profile in mmol/L
triglyceride concentration | 12-months follow-up
  Use of triglyceride concentration to report lipid profile in mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China